CLINICAL TRIAL: NCT02352051
Title: Effects of Atomoxetine and Oros-mph on Executive Functions in Patients With Combined Type Attention Deficit Hyperactivity Disorder
Brief Title: Effects of Atx and Oros-mph on Executive Functions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Bedia İnce Taşdelen, MD, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/580
Record Dates: First submitted 2015-01-14; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Executive Dysfunction
Keywords: attention deficit-hyperactivity disorder (ADHD).; executive functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine group (Active Comparator): The drug was initiated at a dose of 0.5 mg/kg/day which was then gradually increased at 2-week intervals and it was attempted to titrate the dose to 1.2 mg/kg/day.
  Interventions: Drug: Atomoxetine
- Methylphenidate group (Active Comparator): The drug was initiated at the lowest commercially available dose this was then increased at one-month intervals and it was attempted to titrate the dose to 1 mg/kg/day using daily doses of 36-54 mg.
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: Atomoxetine — the drug was initiated at a dose of 0.5 mg/kg/day which was then gradually increased at 2-week intervals and it was attempted to titrate the dose to 1.2 mg/kg/day.
  Other Names: STRATTERA
  Arms: Atomoxetine group
Drug: methylphenidate — the drug was initiated at the lowest commercially available dose this was then increased at one-month intervals and it was attempted to titrate the dose to 1 mg/kg/day using daily doses of 36-54 mg
  Other Names: CONCERTA
  Arms: Methylphenidate group

SUMMARY:
The aim of this study was to evaluate and compare the effects of Atomoxetine(ATX) and osmotic release oral system-methylphenidate (OROS-MPH) therapies on executive functions, activities, treatment response time and adverse effects based on discernible clinical effects in children with combined type attention deficit-hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The aim of this study was to evaluate and compare the effects of Atomoxetine(ATX) and osmotic release oral system-methylphenidate (OROS-MPH) therapies on executive functions, activities, treatment response time and adverse effects based on discernible clinical effects in children with combined type attention deficit-hyperactivity disorder (ADHD).

In this study, the functional capabilities of the patients who clinically responded well to therapy were assessed simultaneously with clinical response that may appear at different time periods and the treatment groups were compared in patients who responded to therapy by excluding patients with insufficient clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Combined type ADHD diagnosis was made by a child psychiatrist according to DSM-IV criteria through K-SADS interview with the patient and mother
* The Clinical Global Impression Scale (CGI-S) was applied to determine ADHD severity and patients with a CGI-S score≥4

Exclusion Criteria:

* Psychological, neurological or psychiatric diseases other than ADHD,
* ADHD types other than combined type,
* Medication that influences cognitive processes or history of such medication,
* WISC-R scores <80 or >120

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Effects of Atx and Oros-mph on Executive Functions, measured by Wisconsin Card Sorting Test, Stroop Test TBAG Form and Visual Auditory Digit Span B | 20 weeks
  Wisconsin Card Sorting Test:WCST measures cognitive processes such as administrative control, characterization, perseveration, executive function, conceptualization, abstract thinking and reasoning, and it is mainly linked to frontal lobe .
  Stroop Test TBAG Form:Stroop test is closely related to frontal lobe and many other serebral regions. It provides information about several cognitive processes such as selective attention, response inhibition, interference control and input processing speed.
  Visual Auditory Digit Span B:VADS B is a test measures short-term memory, sequencing and sensorimotor integration.
  The tests were applied to all patients after diagnosis and evaluations.Recovery score decreasing to 2 or 1 according to CGI-I was set as time for repetition of tests. The tests were repeated at any time of day in ATX group while they were repeated within first 60-180 minutes after ingestion of drug in OROS MPH group.

CONTACTS AND LOCATIONS:
Overall Officials: bedia ince taşdelen, MD, Principal Investigator — TC Erciyes University